CLINICAL TRIAL: NCT06789458
Title: Assessment of Pro-Resolution Mediator Levels in Periodontitis Stage III and IV Before and After Periodontal Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Husam Ghazi Dwerj Alharbi, Husam Ghazi Dwerj Alharbi, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20042024PER7_2_2
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Peridontal Disease
Keywords: lipoxin; proresolution mediators

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Control (No Intervention): Systemically healthy patient
- Periodontitis Stage III and IV (Active Comparator): Professional mechanical plaque control
  Interventions: Procedure: Professional mechanical plaque control

INTERVENTIONS:
Procedure: Professional mechanical plaque control — thisThe first step in therapy is aimed at guiding behavior change by motivating the patient to undertake successful removal of supragingival dental biofilm and risk factor control and may include the following interventions:
  * Interventions to improve the effectiveness of oral hygiene [motivation, instructions (oral hygiene instructions, OHI)
  * Professional mechanical plaque removal (PMPR), which includes the professional interventions aimed at removing supragingival plaque and calculus, as well as possible plaque-retentive factors that impair oral hygiene practices.
  * Adjustment of faulty restoration and polishing
  * The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques.
  Arms: Periodontitis Stage III and IV

SUMMARY:
This study aims to assess Pro-Resolution Mediator levels during non-surgical periodontal therapy in individuals with Stage III and IV periodontitis, comparing them to healthy subjects. Periodontitis, a chronic inflammatory condition affecting tooth-supporting tissues, can lead to tooth loss and systemic complications. Understanding the role of pro-resolving lipid mediators in inflammation resolution may offer insights into therapeutic benefits associated with these mediators.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease that affects the tooth-supporting tissues, it produces a slow destruction of the periodontium that may eventually result in tooth loss. Periodontitis is caused by a dysbiosis of the immune system where there is an imbalance between the processes that activate and terminate the inflammatory process.(Van Dyke, 2020) Pro-resolving lipid mediators (PMs) play a key role in actively resolving inflammation, modulating immune responses, and promoting tissue healing. However, the understanding of PMs in periodontitis and their role in the enduring nature of the disease has not been sufficiently studied in a clinical setting. It has been suggested that PM levels vary between periodontitis patients and healthy individual with periodontal therapy potentially restoring the balance between pro- and anti-inflammatory mediators. (Van Dyke, 2017) The study aims to provide insights into inflammation resolution mechanisms in periodontitis and the therapeutic potential of PMs.

This study aims to Assess Pro-Resolution Mediator Levels During Periodontal Therapy in Patients with Periodontitis Stage III and IV compared to healthy patients.

Hypothesis Null Hypothesis: pro-resolution mediators' level before and after non-surgical treatment in stage III and IV periodontitis compared to healthy patients, there will be no difference in level before and after non-surgical treatment between stage III and IV periodontitis compared to healthy patients.

Trial design:

The current study design is a before and after trial with a single (interventional) population measured before and after treatment compared to a negative control of healthy patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. Adult patients above 18 years old.
2. Interdental CAL at site of greatest loss ≥5 mm or extending to middle third of the root.
3. Interdental CAL at site of greatest loss ≥8 mm or extending to apical third of the root.
4. Probing depth ≥6 mm.
5. Vertical bone loss ≥3 mm.
6. Tooth loss due to periodontitis of ≤4 teeth. (Periodontitis Stage III)
7. Tooth loss due to periodontitis of ≥5 teeth. (Periodontitis Stage IV)
8. Furcation involvement Class II or III Moderate ridge defect.

   -

Exclusion Criteria:

* 1. Pregnancy or lactation. 2. Smoking more than 20 cigarettes. 3. Immuno-inflammatory conditions of the skin and oral mucosa 4. systemic conditions affecting bone turnover and periodontal health status (e.g. endocrine and connective tissue diseases, bisphosphonate antiresorptive therapy, gastrointestinal diseases related to nutrition and mineral metabolism) 5. Periodontal or orthodontic treatment at least 6 months before the start of the study 6. Use of anti-inflammatory and antimicrobial agents within 3 months before sampling

Inclusion criteria for healthy group:

1. Systemically healthy patients.
2. Patients with an age range between 16 to 80 years.
3. Patients have a minimum of 20 teeth.
4. Less than 10% bleeding sites with probing depths ≤3 mm.
5. absence of erythema, oedema.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Change in level of GCF lipoxin A4 | preoperative, one day, one month and 3 months postoperative

SECONDARY OUTCOMES:
Change in level of GCF Protectin | preoperative, one day, one month and 3 months postoperative
Probing pocket depth (PPD) | preoperative, and 3 months postoperative
Bleeding On Probing (BOP) | preoperative, and 3 months postoperative
Plaque index (PI) | preoperative, and 3 months postoperative
Clinical Attachment Level (CAL) | preoperative, and 3 months postoperative
Number of pockets closed | preoperative, and 3 months postoperative

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Dentistry-Cairo University, Manial, Cairo Governorate
  - faculty of dentistry Cairo university, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1186/s12903-024-03948-w